CLINICAL TRIAL: NCT04479059
Title: Endometrial Follicular Fluid Flushing and IVF Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Faik Uzun, research assistant, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ebru Cogendez
Record Dates: First submitted 2020-03-12; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Clinical Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntracavitary fluid flushing (Experimental)
  Interventions: Other: follicular fluid flushing
- Control group (No Intervention)

INTERVENTIONS:
Other: follicular fluid flushing — Follicular fluid obtained during OPU will be used for endometrial cavity flushing.
  Arms: İntracavitary fluid flushing

SUMMARY:
Objective: In this study, our aim will be investigating the pregnancy results in unexplained infertile women undergoing ICSI, by flushing the endometrial cavity with folliculer fluid, that we maintain mature follicules inside them in oocyte retrieval day.

Study Design: 100 subfertile women who applied to Zeynep Kamil Hospital, In Vitro Fertilization Center between October 2016 to May 2017 will be randomized with computer generated programme. The patients will be divided into two groups; follicular fluid group (n=50) and control group (n=50). The inclusion criterias are: age between 20-39 years, basal FSH level < 10 mIU/ml, body mass index<35 kg/m2 and E2 levels in human chorionic gonadotropin (hCG) day between 1000-4000 pg/ml. Patients meets these criteria will be included to the study programme. The exclusion criteria are determined as below: previously diagnosed endometriosis, uterine leiomyomas, hydrosalpinx, endocrinological disorders; previous history of implantation failure in IVF/ICSI cycles and severe male factor infertility.

DETAILED DESCRIPTION:
Objective: In this study, our aim will be investigating the pregnancy results in unexplained infertile women undergoing ICSI, by flushing the endometrial cavity with folliculer fluid, that we maintain mature follicules inside them in oocyte retrieval day.

Study Design: 100 subfertile women who applied to Zeynep Kamil Hospital, In Vitro Fertilization Center between October 2016 to May 2017 will be randomized with computer generated programme. The patients will be divided into two groups; follicular fluid group (n=50) and control group (n=50). The inclusion criterias are: age between 20-39 years, basal FSH level < 10 mIU/ml, body mass index<35 kg/m2 and E2 levels in human chorionic gonadotropin (hCG) day between 1000-4000 pg/ml. Patients meets these criteria will be included to the study programme. The exclusion criteria are determined as below: previously diagnosed endometriosis, uterine leiomyomas, hydrosalpinx, endocrinological disorders; previous history of implantation failure in IVF/ICSI cycles and severe male factor infertility.

ELIGIBILITY:
inclusion criteria:age between 20-39 years, basal FSH level < 10 mIU/ml, body mass index<35 kg/m2 and E2 levels in human chorionic gonadotropin (hCG) day between 1000-4000 pg/ml. -

Exclusion Criteria:previously diagnosed endometriosis, uterine leiomyomas, hydrosalpinx, endocrinological disorders; previous history of implantation failure in IVF/ICSI cycles and severe male factor infertility.

-

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — infertile women
Enrollment: 100 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | during last 24 months
  intrauterine pregnancy with metal cardiac activity

IPD SHARING:
Plan to Share IPD: No